CLINICAL TRIAL: NCT01011062
Title: Effect of Acute Angiotensin Receptor Blockade on Insulin Resistance and Selected Cytokines in Adipose Tissue in Type 2 Diabetes
Brief Title: Effect of Angiotensin Receptor Blockade on Insulin Resistance and Adipose Tissue Cytokines in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Dagmar Köveslygetyova, Diabetes Center, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CDS01
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2009-11

CONDITIONS: Insulin Resistance; Type 2 Diabetes
Keywords: Adipose tissue; Adipokines
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Losartan; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hyperinsulinaemia (Experimental): Hyperinsulinaemic (1 mIU/kg/min) euglycaemic (5 mmol/l) clamp
  Interventions: Procedure: Hyperinsulinaemia
- Losartan + hyperinsulinaemia (Experimental)
  Interventions: Procedure: Hyperinsulinaemia; Drug: Losartan
- Saline (Placebo Comparator): Infusion of Saline as a volume control intervention
  Interventions: Drug: Saline

INTERVENTIONS:
Procedure: Hyperinsulinaemia — Hyperinsulinaemic (1 mIU/kg/min) euglycaemic (5 mmol/l) clamp
  Arms: Hyperinsulinaemia; Losartan + hyperinsulinaemia
Drug: Losartan — Acute administration of losartan 200mg total prior to clamp
  Arms: Losartan + hyperinsulinaemia
Drug: Saline — Infusion of Saline as a volume control intervention
  Arms: Saline

SUMMARY:
The study aims to investigate the effect of acute angiotensin receptor blockade on insulin action/insulin resistance and expressions of selected adipocytokines in subcutaneous adipose tissue in insulin-resistant subjects with type 2 diabetes and healthy controls.

Hypothesis: Changes in adipocytokine concentrations and/or expressions and different reactions to acute in vivo induced hyperinsulinemia and angiotensin receptor blockade will be found in patients with type 2 diabetes compared to healthy subjects. A significant relationships between insulin sensitivity and selected adipokines and intracellular fat content and high energy phosphates in soleus muscle will be documented in healthy individuals, while no significant relation will be found in patients with type 2 diabetes.

DETAILED DESCRIPTION:
10-15 patients with type 2 diabetes and 10-15 healthy control subjects will be examined on an outpatient basis. The following examination will be carried out in each subject after 12 hrs fasting:

* Oral glucose tolerance test (75 g of glucose) (in healthy subjects to confirm the normal tolerance of glucose).
* Evaluation of insulin secretion after 1 mg of glucagon i.v.
* Hyperinsulinaemic (75 milly-international unit(mIU)/l) euglycemic clamp study lasting 4 hours combined with indirect calorimetry and biopsy of subcutaneous adipose tissue.
* Hyperinsulinemic (75 mIU/l) euglycemic clamp study lasting 4 hours combined with indirect calorimetry after losartan 100 mg given in the evening and in the morning before the study.
* Proton and phosphorus magnetic resonance spectroscopy.

Before (0 min), at 30 min and in the end of studies c) and d) the blood samples will be taken and biopsies of subcutaneous abdominal adipose tissue will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 Diabetes treated with oral agents and/or diet
2. Healthy volunteers age- and sex-matched to type 2 diabetes, without any concomitant disease

Exclusion Criteria:

1. Type 2 Diabetes

   * treated with insulin
   * clinical evidence of atherosclerotic complications
   * advanced long-term diabetic complications (manifest nephropathy, proliferative retinopathy)
   * other internal disease
   * weight change >10% 3 months prior to study
2. Healthy volunteers

   * fulfilling the criteria of metabolic syndrome
   * weight change >10% 3 months prior to study

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity measured as glucose disposal during clamp | 4 hours

SECONDARY OUTCOMES:
plasma adipokines and their expressions in SAT | at 0 and 240 min of the clamp

CONTACTS AND LOCATIONS:
Overall Officials: Terezie Pelikanova, Prof., MD, Principal Investigator — Diabetes Center, Institute of Clinical and Experimental Medicine
Locations (1):
- Diabetes Center, Institute of Clinical and Experimental Medicine, Prague, Czechia